CLINICAL TRIAL: NCT04867811
Title: Effect of Transcutaneous Electrical Nerve Stimulation and Cupping Therapy in The Treatment of Tennis Elbow: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Emad Eldin Mohamed, lecturer, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7645
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Tennis Elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Cupping Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group A (Experimental): received conventional therapy
  Interventions: Other: conventional therapy
- group B (Experimental): received TENS in addition to conventional therapy
  Interventions: Other: conventional therapy; Device: TENS
- group C (Experimental): received cupping therapy with conventional therapy
  Interventions: Other: conventional therapy; Other: cupping therapy
- group D (Experimental): TENS and cupping therapy plus conventional therapy
  Interventions: Other: conventional therapy; Other: TENS and cupping therapy

INTERVENTIONS:
Other: conventional therapy — conventional therapy
Other: cupping therapy — cupping therapy
  Arms: group C
Device: TENS — transcutaneous electrical nerve stimulation
  Arms: group B
Other: TENS and cupping therapy — TENS and cupping therapy
  Arms: group D

SUMMARY:
One hundred and twenty patients (67 females and 53 males) with unilateral TE were included in the study from January 2020 to December 2020 and diagnosed by an orthopedist. Their ages ranged between 20 and 50 years old.

DETAILED DESCRIPTION:
They were divided randomly into three groups by lottery method. Group A (n=30) received conventional therapy, group B (n=30) received TENS in addition to conventional therapy, group C received cupping therapy with conventional therapy and group D (n=30) received TENS and cupping therapy plus conventional therapy. All patients read and signed a consent form before participation in this trial. This study was approved by the Ethical Committee of the Faculty of Physical Therapy, October 6 University, Egypt. Patients with pain in the lateral epicondylar region, increased pain with pressure and resistance to wrist extension, persistence of symptoms for more than three months, no physical therapy interventions during the last three months were included in the study while patients with bilateral tennis elbow, proximal radio-ulnar joint synovitis, radial nerve entrapment, cervical spine radiculopathy, other diseases like medial epicondylitis, impaired sensibility and paralysis that may affect the outcome measurement and previous injury or surgery in the region of common extensor origin were excluded from this study.

ELIGIBILITY:
Inclusion Criteria:

- Patients with pain in the lateral epicondylar region, increased pain with pressure and resistance to wrist extension, persistence of symptoms for more than three months, no physical therapy interventions during the last three months

Exclusion Criteria:

* patients with bilateral tennis elbow, proximal radio-ulnar joint synovitis, radial nerve entrapment, cervical spine radiculopathy, other diseases like medial epicondylitis, impaired sensibility and paralysis that may affect the outcome measurement and previous injury or surgery in the region of common extensor origin

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-12 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 weeks
Pain-Free Grip Strength | 4 weeks
Patient-Rated Tennis Elbow Evaluation (PRTEE) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Bassam, Qaliubia, Egypt

IPD SHARING:
Plan to Share IPD: No